CLINICAL TRIAL: NCT06276348
Title: Newborn Genomic Sequencing (BeginNGS) Prospective Pilot Study
Brief Title: Newborn Genomic Sequencing Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rady Pediatric Genomics & Systems Medicine Institute (Other)
Responsible Party: Principal Investigator, Stephen F. Kingsmore, President and CEO, Rady Pediatric Genomics & Systems Medicine Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 20226892
Record Dates: First submitted 2024-02-16; First posted 2024-02-26 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Genetic Disease
MeSH Terms: conditions — Genetic Diseases, Inborn | interventions — Whole Genome Sequencing

STUDY DESIGN:
Intervention Model Description: Single group, multiple interventions. All enrollees receive all interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enrollees (Experimental): Enrolled infants will receive 3 tests (DWGS, BeginNGS, and WES). DWGS will be performed in a standard manner. BeginNGS and WES will be performed in a batch after completion of enrollment. The diagnostic sensitivity and specificity of BeginNGS and WES will be compared to DWGS (a standard clinical test compliant with the Clinical Laboratory Improvement Amendments Act).
  Interventions: Genetic: Whole genome sequencing; Genetic: BeginNGS test; Genetic: WES

INTERVENTIONS:
Genetic: Whole genome sequencing — Standard diagnostic whole genome sequencing will be performed.
Genetic: BeginNGS test — Genomic sequencing that screens for 434 genetic diseases.
Genetic: WES — Whole exome sequencing will be performed.

SUMMARY:
The goal of this clinical trial is to test a new method for newborn screening using whole genome sequencing, called BeginNGS. Newborns who are not suspected of having genetic diseases and who are admitted to the NICU at Rady Children's Hospital, San Diego, will be enrolled. The main questions this study aims to answer are:

* What is the diagnostic yield of diagnostic whole genome sequencing (DWGS) in this population?
* What is the diagnostic sensitivity and specificity of BeginNGS and whole exome sequencing (WES) as compared to DWGS?
* What are the potential issues related to implementing DWGS in this population?

Enrolled newborns will have a blood sample taken and will receive three tests:

* DWGS
* BeginNGS
* WES

DETAILED DESCRIPTION:
Newborn screening (NBS) by testing dried blood spots (DBS) identifies newborns with a few diseases for which effective treatments are available to enable treatment at or before symptom onset. Because NBS improves outcomes in these diseases, it is performed on almost all US babies. The current Federal recommended NBS list is limited to 35 conditions and identifies ~6,600 affected children per year. In genetic diseases not screened by NBS, however, outcomes remain poor because of delays in diagnosis and treatment. The investigators recently developed a system for NBS for 434 severe, childhood genetic diseases for which effective treatments are available using whole genome sequencing (WGS), called BeginNGS. Retrospective studies showed BeginNGS to have a true negative rate (specificity) of 99.7% and true positive rate (sensitivity) of 88.8%. The investigators now propose to undertake a first prospective study in newborns admitted to the Neonatal Intensive Care Unit (NICU) at Rady Children's Hospital, San Diego (RCHSD) to compare the sensitivity and specificity of BeginNGS with that of standard, diagnostic rapid whole genome sequencing (DWGS) and whole exome sequencing (WES). This study is in preparation for larger, future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Neonates less than or equal to 10 days old who are admitted to the RCHSD NICU.

Exclusion Criteria:

1. Neonates who have enrolled in another clinical study at Rady Children's Institute for Genomic Medicine or in whom DWGS has been ordered or is being considered.
2. Neonates whose mother is less than 18 years of age.
3. Neonates who are wards of the state.
4. Neonates whose parent/legal guardian is unable to provide consent.

Ages: 1 Day to 10 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Proportion of enrolled infants who are diagnosed with a genetic disease by DWGS. | 18 months
  Proportion

SECONDARY OUTCOMES:
Proportion of enrolled infants who are identified with a genetic disease by BeginNGS. | 18 months
  Proportion
Proportion of enrolled infants who are identified with a genetic disease by WES. | 18 months
  Proportion
Proportion of enrolled infants who have a positive standard NBS test. | 18 months
  Proportion
Proportion of parents approached who agree to participate in the study. | 18 months
  Proportion
Parental reasons for refusal. | 18 months
  Questionnaire
Time from sample arriving in lab to return of DWGS results. | 18 months
  Time (days)
Time from birth to return of DWGS results. | 18 months
  Time (days)
Results of confirmatory testing if BeginNGS or WES identifies a diagnostic finding not reported by DWGS. | 18 months
  Proportion of findings confirmed

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Kingsmore, MD DSc, Principal Investigator — Rady Children's Institute for Genomic Medicine
Locations (1):
- Rady Children's Hospital San Diego, San Diego, California, United States